CLINICAL TRIAL: NCT07104968
Title: Mild and Moderate Aortic Regurgitation: Risk Factors for Progress and Outcome
Status: Not yet recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Region Västmanland (Other)
Responsible Party: Principal Investigator, Pär Hedberg, Associate professor, Region Västmanland
Other Study IDs: 2025-02671-01
Record Dates: First submitted 2025-07-25; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Aortic Regurgitation
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with aortic regurgitation: Observational study, no interventions

SUMMARY:
This observational study aims to evaluate risk factors of progress and adverse outcome of aortic regurgitation

DETAILED DESCRIPTION:
Aortic regurgitation is relatively common, with a prevalence of 13% for men and 8,5% for women in the Framingham study (Singh et al). Patients with aortic regurgitation are evaluated regularly with echocardiography to see if progress occurs, and suitable candidates are referred for surgical repair or replacement of the aortic valve.

However, an American study from 2019 showed that only 12% of cases of aortic regurgitation progressed from mild to moderate or severe over a 10 years period (Yang et al). This means that the majority of patients undergo echocardiographic evaluations without a clinical benefit.

It is unclear whether these findings also apply to a Swedish population with the European definitions for aortic regurgitation.

Aim:

To do a retrospective analysis of patients evaluated with echocardiography in Västerås, Sweden between January 2003 and March 2025 to describe the prevalence of aortic regurgitation as well as aortic dilatation, to describe how often progress occurs in patients with mild or moderate aortic regurgitation, and finally to look at factors (clinical, echocardiographic) associated with progress of aortic regurgitation as well as outcome (mortality, MACE, cardiac surgery).

ELIGIBILITY:
Inclusion Criteria:

* Patients investigated with echocardiography between January 2003 and March 2025
* Age ≥18 years
* At least minimal aortic regurgitation
* At least one additional echocardiography after the index investigation

Exclusion Criteria:

* Age <18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with aortic regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 35000 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Progress of aortic regurgitation | Depending on when the patients was evaluated first, up to approximately 20 years of follow-up
  Progress of aortic regurgitation from mild to moderate or severe, or moderate to severe. Progress is defined according to current European Society for Cardiology guidelines using a comprehensive echocardiographic assessment

SECONDARY OUTCOMES:
Surgical treatment of aortic regurgitation or aortic aneurysm | Depending on when the patients was evaluated first, up to approximately 20 years of follow-up
  Surgical treatment of aortic regurgitation or aortic aneurysm
Hospitalization for heart failure | Depending on when the patients was evaluated first, up to approximately 20 years of follow-up
  Hospitalization for heart failure during follow-up
Hospitalization for stroke or myocardial infarction | Depending on when the patients was evaluated first, up to approximately 20 years of follow-up
  Composite endpoint
All-cause mortality | Depending on when the patients was evaluated first, up to approximately 20 years of follow-up
  All-cause mortality during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Matthijs Velders, MD PhD, Principal Investigator — Region Västmanland
Locations (1):
- Västmanlands sjukhus Västerås, Västerås, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yang LT, Enriquez-Sarano M, Michelena HI, Nkomo VT, Scott CG, Bailey KR, Oguz D, Wajih Ullah M, Pellikka PA. Predictors of Progression in Patients With Stage B Aortic Regurgitation. J Am Coll Cardiol. 2019 Nov 19;74(20):2480-2492. doi: 10.1016/j.jacc.2019.08.1058. PMID 31727286
- [Background] Singh JP, Evans JC, Levy D, Larson MG, Freed LA, Fuller DL, Lehman B, Benjamin EJ. Prevalence and clinical determinants of mitral, tricuspid, and aortic regurgitation (the Framingham Heart Study). Am J Cardiol. 1999 Mar 15;83(6):897-902. doi: 10.1016/s0002-9149(98)01064-9. PMID 10190406